CLINICAL TRIAL: NCT00418054
Title: Phase II, Multi-Center, Randomized, Double-Blind Study of Nitazoxanide Tablets Combined With Peginterferon Compared to Peginterferon Monotherapy in the Treatment of Chronic Hepatitis C
Brief Title: Study of Nitazoxanide Combined With Peginterferon Compared to Peginterferon Monotherapy in the Treatment of Hepatitis C
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Romark Laboratories L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RM01-2022
Record Dates: First submitted 2007-01-03; First posted 2007-01-04 (Estimated); Last update posted 2007-01-04 (Estimated); Status verified 2007-01

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — nitazoxanide; peginterferon alfa-2b

INTERVENTIONS:
Drug: Nitazoxanide plus peginterferon alfa-2b
Drug: Peginterferon alfa-2b

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of nitazoxanide-peginterferon alfa-2b combination therapy compared to peginterferon monotherapy in patients that are treatment naive or pre-treated for 24 weeks with nitazoxanide monotherapy in the treatment of chronic hepatitis C.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Chronic hepatitis C infection (at least 6 months) evidenced by a positive enzyme immunoassay for anti-HCV-antibodies and a positive quantitative RT-PCR amplification of HCV RNA.
* Chronic inflammation on liver biopsy compatible with a diagnosis of chronic viral hepatitis.
* HCV genotype 4.
* Patients that have not previously received peginterferon.

Exclusion Criteria:

* Patients unable to take oral medications.
* Use of ribavirin within 30 days prior to enrollment.
* Females who are either pregnant, breast-feeding or not using birth control and are sexually active.
* Any investigational drug therapy within 30 days prior to enrollment other than through Romark study number RM01-3027.
* Patients with other causes of liver disease.
* Transplant recipients receiving immune suppression therapy.
* Patient co-infected with human immunodeficiency virus, hepatitis A virus, hepatitis B virus, or hepatitis D virus based on enzyme immunoassay.
* Patients with decompensated cirrhosis, thrombocytopenia (platelet count <80,000), neutropenia, history of variceal bleeding, ascites, hepatic encephalopathy or CTP scores >6.
* Patients with history of alcoholism (unless abstinent for 2 years) or with an alcohol consumption of >20 grams per day.
* Patients who are clinically unstable.
* Patients with any concomitant condition that, in the opinion of the investigator would preclude evaluation of response or make it unlikely that the contemplated course of therapy and follow-up could be completed.
* History of hypersensitivity or intolerance to any of the excipients comprising the nitazoxanide tablets or peginterferon alfa-2b solution for injection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2005-12; Study Completion 2006-07

PRIMARY OUTCOMES:
Virologic response

SECONDARY OUTCOMES:
2 log drop in serum HCV RNA
Change in ALT

CONTACTS AND LOCATIONS:
Overall Officials: Yehia El-Gohary, MD, Principal Investigator — Department of Tropical Medicine & Infectious Diseases, Alexandria University; Asem Elfert, MD, Principal Investigator — Department of Tropical Medicine & Infectious Diseases, Tanta University School of Medicine
Locations (2):
- Egypt (2):
  - Department of Tropical Medicine & Infectious Diseases, Alexandria University, Alexandria
  - Department of Tropical Medicine & Infectious Diseases, Tanta University School of Medicine, Tanta